CLINICAL TRIAL: NCT00861263
Title: The Clinical Utility of Overtube Use at the Time of Endoscopy
Acronym: Spirus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Spirus Overtube
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Small Bowel Visualization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- spiral overtube (Other): Any subject that has been referred for spiral enteroscopy will be asked to participate in this study. The purpose is to gather data about the technical aspects of the procedure,diagnostic capability and treatment as well as long term follow up.
  Interventions: Device: overtube use during enteroscopy

INTERVENTIONS:
Device: overtube use during enteroscopy — use of overtube for the regular scheduled enteroscopy

SUMMARY:
Endoscopy has become a vital part of the gastroenterologist's evaluation and treatment of disorders involving the gastrointestinal (GI) tract. The small bowel is an area of the GI tract, which can prove difficult to visualize during an endoscopy specifically designed to evaluate it, termed enteroscopy. Thus, the FDA has approved overtubes, such as the Endo-Ease® spiral overtube (Spirus Medical, Inc.) or EnteroPro® balloon overtube (Olympus Medical, Inc.), to facilitate passage of the endoscope through the GI tract. The aims of the study are to evaluate the efficiency of an overtube system for visualization of small bowel. The hypothesis is that this will permit more complete and efficient evaluation of the small intestine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years.
2. Have an indication for enteroscopy as determined by the patient's physicians. These indications include, but are not limited to, obscure gastrointestinal bleeding, malabsorption, suspected small bowel tumor, small bowel strictures, small bowel ulceration, and abnormal imaging of the small bowel.
3. Scheduled to undergo enteroscopy at the University of Florida, Gainesville, Florida, as medically indicated.
4. Subject must be able to give informed consent.

Exclusion Criteria:

1. Platelets < 75,000.
2. INR > 1.6.
3. NSAIDS within 48 hours of procedure.
4. Pregnancy.
5. Esophageal stricture.
6. Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2007-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida, Division of Gastroenterology
Locations (1):
- Shands at UF, Gainesville, Florida, United States

REFERENCES:
- [Derived] Williamson JB, Judah JR, Gaidos JK, Collins DP, Wagh MS, Chauhan SS, Zoeb S, Buscaglia JM, Yan H, Hou W, Draganov PV. Prospective evaluation of the long-term outcomes after deep small-bowel spiral enteroscopy in patients with obscure GI bleeding. Gastrointest Endosc. 2012 Oct;76(4):771-8. doi: 10.1016/j.gie.2012.05.025. Epub 2012 Jul 7. PMID 22771101
- [Derived] Judah JR, Collins D, Gaidos JK, Hou W, Forsmark CE, Draganov PV. Prospective evaluation of gastroenterologist-guided, nurse-administered standard sedation for spiral deep small bowel enteroscopy. Dig Dis Sci. 2010 Sep;55(9):2584-91. doi: 10.1007/s10620-010-1335-x. Epub 2010 Jul 15. PMID 20632098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We started this study in June 2007 and ended this study in Oct 2012. We approached any patient who was scheduled in our endoscopy suite for an overtube enteroscopy.
Pre-assignment Details: The only significant event was that the subject was scheduled for an enteroscopy in our facility and a overtube was used at the time of endoscopy.
Groups:
- Enteroscopy: Any subject who was referred for an enteroscopy to our facility and an overtube was used at the time of endoscopy was asked to participate in this study.
Period: Overall Study
Arm/Group | Enteroscopy
Started | 193
Completed | 193
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enteroscopy
Number analyzed (Participants) | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 94
  >=65 years | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 92
Region of Enrollment [Number; unit: participants]
  United States | 193

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Persistent or Recurrent Bleeding
Description: The number of patients that had persistent or recurrent GI bleeding after spiral enteroscopy.
Time Frame: up to 6 yrs after after the endoscopy
Measure: Number; unit: participants
Groups:
- Spiral Enteroscopy Subjects: All subjects followed up after spiral enteroscopy
Arm/Group | Spiral Enteroscopy Subjects
Number analyzed (Participants) | 61
participants | 16 (12.3)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected for 6 years.
Arm/Group | Enteroscopy
Serious Adverse Events (participants affected / at risk) | 8/193
Other Adverse Events (participants affected / at risk) | 0/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enteroscopy (N=193)
Bradycardia (Cardiac disorders) | 2 (2) — Two subjects experienced bradycardias during endoscopy and were hospitalized overnight for observation.
Chest pain (Cardiac disorders) | 1 (1) — One subject experience Chest pain after endoscopy and was hospitalized overnight for observation.
Transient Ischemic Attack (Vascular disorders) | 1 (1) — One subject experienced a transient ischemic attack after endoscopy and was hospitalized overnight for observation.
Ventrical Tachycardia Arrest (Cardiac disorders) | 1 (1) — One subject experienced a ventrical tachycardia arrest and was hospitalized.
Partial Thickness Mucosal Tear (Gastrointestinal disorders) | 3 (3) — Three subjects experienced a partial thickness mucosal tear as part of their endoscopy.

LIMITATIONS AND CAVEATS:
No limitations were found

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No